CLINICAL TRIAL: NCT03741049
Title: Evaluation of the Novel ScalpelCric Set for Cricothyrotomy Corresponding the Scalpel-Bougie Technique and Comparison With Two Further Techniques of Cricothyrotomy on a Plastic Laryngeal Model (A) and Comparison of the Novel ScalpelCric Set With Surgical Cricothyrotomy in a Porcine Laryngeal Model (B) Influence of Training (A+B) in a Simulation
Brief Title: Evaluation of the ScalpelCric Set and Comparison With Two Further Techniques of Cricothyrotomy
Status: Completed | Type: Observational
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Nina Pirlich, Dr. med., Principal Investigator, Johannes Gutenberg University Mainz
Other Study IDs: 2018-13819
Record Dates: First submitted 2018-11-08; First posted 2018-11-14 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Cricothyroidotomy
Keywords: CVCI; Emergency medicine; Airway management; Cricothyroidotomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Consultants
  Interventions: Device: Scalpel Bougie technique (plastic laryngeal model); Device: Seldinger technique (plastic laryngeal model); Device: Surgical technique (plastic laryngeal model); Device: Scalpel Bougie technique (porcine laryngeal model); Device: Surgical technique (porcine laryngeal model)
- Trainee anaesthetists
  Interventions: Device: Scalpel Bougie technique (plastic laryngeal model); Device: Seldinger technique (plastic laryngeal model); Device: Surgical technique (plastic laryngeal model); Device: Scalpel Bougie technique (porcine laryngeal model); Device: Surgical technique (porcine laryngeal model)
- Paramedics
  Interventions: Device: Scalpel Bougie technique (plastic laryngeal model); Device: Seldinger technique (plastic laryngeal model); Device: Surgical technique (plastic laryngeal model)
- Students
  Interventions: Device: Scalpel Bougie technique (plastic laryngeal model); Device: Seldinger technique (plastic laryngeal model); Device: Surgical technique (plastic laryngeal model)

INTERVENTIONS:
Device: Scalpel Bougie technique (plastic laryngeal model) — ScalpelBougie Set
Device: Seldinger technique (plastic laryngeal model) — Melker Set
Device: Surgical technique (plastic laryngeal model) — Scalpel and speculum
Device: Scalpel Bougie technique (porcine laryngeal model) — ScalpelCric Set
  Groups: Consultants; Trainee anaesthetists
Device: Surgical technique (porcine laryngeal model) — Scalpel and speculum
  Groups: Consultants; Trainee anaesthetists

SUMMARY:
During a cannot ventilate cannot intubate situation surgical airway is the last rescue option. Especially in the prehospital setting the airway management seems to be more difficult than in a hospital setting. Nearly all emergency physicians have a limited experience with cricothyrotomy and it is a unclear what method should be taught for this lifesaving procedure, due to lack of data in humans. The aim of this study is to compare the performance of medical personnel (medical students, paramedics, trainee anaesthetists and consultants) in establishing an emergency surgical airway on a plastic laryngeal model and in a porcine laryngeal model using the Scalpel Bougie technique, the Seldinger technique and the common surgical technique.

Furthermore the investigators want to elucidate whether the training of the 3 techniques has an influence in the decision making of the preferred technique in a subsequently simulated cannot ventilate cannot intubate scenario.

DETAILED DESCRIPTION:
The investigators plan to recruit medical students (University Mainz), paramedics (employed in ambulance and rescue helicopter), trainee anaesthetists and consultants of the department of anesthesiology from the university hospital Mainz. After written informed consent the participants have to complete an pre-study questionnaire, than the participants get an information sheet about the 3 techniques and the investigators show the participants a short video demonstrating the different techniques. All participants have the opportunity to practice one insertion with each method on a plastic laryngeal model.

After that the participants have to perform each technique on the plastic model and the investigators measure the time from initially handling equipment to the final end-point, which the investigators take as a successful placement of the endotracheal tube verified by a fiberoptic position check.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* German language in speaking and writing
* Capability of giving consent

Exclusion Criteria:

* Participants unwilling or unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Medical students (University Mainz), paramedics (DRK, MHD, ASB, ADAC), trainee anaesthetists and consultants (Department of anaesthesiology University hospital Mainz)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2018-11-13 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2018-12-20 (Actual)

PRIMARY OUTCOMES:
Time from initially handling equipment to a successful placement of the endotracheal tube verified by a fiberoptic position check | up to 3 minutes

SECONDARY OUTCOMES:
Success rate in the first trial | up to 3 minutes
Number of trials | up to 3 minutes
Dimension of the tracheal trauma | up to 10 minutes
  horizontally and vertically in mm
Comfort evaluation by the performer | up to 15 minutes
  Likert-Scale: 1=very easy, 2=easy, 3=difficult, 4=very difficult
Influence of training on the time to decision making for cricothyrotomy | up to 5 hours
  After performing the different techniques of cricothyrotomy on a platistic and a porcine laryngeal model, the participants will complete a simulator training for a cannot intubate and cannot ventilate scenario. Time to decide (measured in seconds) to perform cricothyrotomy will be measured from the beginning of the scenario.
Influence of training on choosing the technique | up to 5 hours
  After performing the different techniques of cricothyrotomy on a platistic and a porcine laryngeal model, the participants will complete a simulator training for a cannot intubate and cannot ventilate scenario. The technique (Scalpel bougie, seldinger, surgical) of cricotyrotomy, chosen by the participant will be reported and compared with the preferred technique, the participant had chosen before performing the training.

CONTACTS AND LOCATIONS:
Locations (1):
- Johannes Gutenberg University Medicine Centre Mainz, Mainz, Rhineland Palatine, Germany